CLINICAL TRIAL: NCT04014725
Title: Validation of the Utility of Myopia Intelligent Diagnostic System: A Clinical Trial
Brief Title: Validation of the Utility of Myopia Intelligent Diagnostic System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CCPMOH2019-China-2
Record Dates: First submitted 2019-07-01; First posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eligible patients for AI test (Experimental)
  Interventions: Device: Myopia Intelligent Diagnostic System

INTERVENTIONS:
Device: Myopia Intelligent Diagnostic System — An artificial intelligence to make diagnosis of myopia using ocular appearance images

SUMMARY:
The screening of myopia via artificial intelligence represents an challenge in computational medicine. Here, the investigators use "deep learning" to create an automatic diagnostic system for myopia screening using ocular appearance images. The investigator also use this system and conduct clinical trial to validate its performance.

ELIGIBILITY:
Inclusion Criteria:

* Student aged 6-18

Exclusion Criteria:

-

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-07-10 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
The AUC of the Myopia Intelligent Diagnostic System | up to 3 month

SECONDARY OUTCOMES:
The sensitivity of the Myopia Intelligent Diagnostic System | up to 3 month
The specificity of the Myopia Intelligent Diagnostic System | up to 3 month